CLINICAL TRIAL: NCT01178866
Title: Markers of Tissue Perfusion as Predictors of Complicated Evolution in Patients With Left Ventricular Dysfunction Submitted to Coronary Artery Bypass Surgery
Brief Title: Laboratory Outcome Predictors in Coronary Surgery
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Thiana Yamaguti/ Médica assistente da divisão de anestesiologia do InCor - HCFMUSP, University of Sao Paulo
Other Study IDs: HC517/04
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2008-01

CONDITIONS: Left Ventricular Dysfunction; Coronary Artery Bypass Surgery; Tissue Hypoperfusion
Keywords: thoracic surgery; myocardial revascularization; left ventricular dysfunction; tissue perfusion; prognosis
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clinical course: complicated course group (death within 30 days after surgery or ICU stay > 4 days) and uncomplicated course group (ICU stay ≤ 4 days).

SUMMARY:
Evaluate less employed markers of tissue hypoperfusion as venoarterial carbon dioxide partial pressure difference (ΔPCO2) and estimated respiratory quotient (eRQ) combined to other classically studied markers as predictive factors of complicated clinical course after cardiac surgery in patients with left ventricular dysfunction.

DETAILED DESCRIPTION:
Patients with left ventricular dysfunction are more susceptible to tissue hypoperfusion and presents more frequently both low cardiac output syndrome and systemic inflammatory response, what results in prolonged stay in intensive care unit (ICU), and higher mortality rates when compared to patients with normal ventricular function.

The early prediction of prolonged ICU stay through the detection of tissue hypoperfusion may improve the management of care and decrease morbidity of this particular group of patients. However, classic markers of tissue hypoxia as central venous saturation, base excess, lactate may not be predictors of outcome in cardiac surgery patients with left ventricular dysfunction.

The question addressed in this study is if less employed markers of tissue hypoperfusion as as venoarterial carbon dioxide partial pressure difference (ΔPCO2) and estimated respiratory quotient (eRQ) have predictive value of prolonged ICU stay in patients with left ventricular dysfunction submitted to coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults
* left ventricular dysfunction (ejection fraction < 50%)
* patients undergoing coronary artery bypass surgery requiring the use of Cardiopulmonary Bypass (CPB)

Exclusion Criteria:

* renal failure (creatinine clearance lower than 40 ml/min/m2),
* hepatic dysfunction
* endocrinologic disorders
* pulmonary disease
* uncontrolled diabetes mellitus
* a history of fever or infection within the week before surgery
* previous anemia (hemoglobin ≤ 10.0 g/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing coronary artery bypass surgery requiring the use of CPB
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Complicated clinical course after coronary artery bypass surgery | within the first 30 days after surgery
  Complicated clinical course defined as death within the first 30 days after surgery or ICU stay more than 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Thiana Yamaguti, PhD, Principal Investigator — Heart Institute, Hospital of Clinics, São Paulo University Medical School; José Otávio C. Auler Júnior, PhD/Chairman, Study Chair — Heart Institute, Hospital of Clinics, São Paulo University Medical School; Marilde A. Piccioni, PhD, Study Director — Heart Institute, Hospital of Clinics, São Paulo University Medical School
Locations (1):
- Heart Institute, Hospital of Clinics, São Paulo University Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Mekontso-Dessap A, Castelain V, Anguel N, Bahloul M, Schauvliege F, Richard C, Teboul JL. Combination of venoarterial PCO2 difference with arteriovenous O2 content difference to detect anaerobic metabolism in patients. Intensive Care Med. 2002 Mar;28(3):272-7. doi: 10.1007/s00134-002-1215-8. Epub 2002 Feb 8. PMID 11904655
- [Background] Ranucci M, De Toffol B, Isgro G, Romitti F, Conti D, Vicentini M. Hyperlactatemia during cardiopulmonary bypass: determinants and impact on postoperative outcome. Crit Care. 2006;10(6):R167. doi: 10.1186/cc5113. PMID 17134504
- [Background] Ranucci M, Isgro G, Romitti F, Mele S, Biagioli B, Giomarelli P. Anaerobic metabolism during cardiopulmonary bypass: predictive value of carbon dioxide derived parameters. Ann Thorac Surg. 2006 Jun;81(6):2189-95. doi: 10.1016/j.athoracsur.2006.01.025. PMID 16731152
- [Background] Meregalli A, Oliveira RP, Friedman G. Occult hypoperfusion is associated with increased mortality in hemodynamically stable, high-risk, surgical patients. Crit Care. 2004 Apr;8(2):R60-5. doi: 10.1186/cc2423. Epub 2004 Jan 12. PMID 15025779
- [Background] Topkara VK, Cheema FH, Kesavaramanujam S, Mercando ML, Cheema AF, Namerow PB, Argenziano M, Naka Y, Oz MC, Esrig BC. Coronary artery bypass grafting in patients with low ejection fraction. Circulation. 2005 Aug 30;112(9 Suppl):I344-50. doi: 10.1161/CIRCULATIONAHA.104.526277. PMID 16159844